CLINICAL TRIAL: NCT03676725
Title: Assessing the Frequency of Lidocaine Ineffectiveness in the General Population vs. Males With ADHD, and Females With ADHD, With or Without PMS
Brief Title: Prevalence of Lidocaine Ineffectiveness in Adults With and Without ADHD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: PhenoSolve, LLC (Industry)
Collaborators: Jacobi Medical Center (Other); Boston Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-272
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: ADHD; PMS
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: A group of 100 subjects will be assessed.
Masking Description: The scoring of the lidocaine test is masked, using the coded identity of the tastes. The tastes will be assessed in random order. The subjects and other study personnel will be told not to discuss what the subject could or couldn't taste. Scoring will not be shared with the testing site until all testing is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All subjects (Experimental): All subjects get the lidocaine taste test
  Interventions: Drug: Lidocaine gel

INTERVENTIONS:
Drug: Lidocaine gel — Lidocaine gel (0.75 g premeasured dose of Septodont 5% oral gel NDC 0362-0221-10)
  Other Names: Intervention

SUMMARY:
This work will assess the prevalence in the general population of the ineffectiveness of the anesthetic Lidocaine compared to males with ADHD and females with ADHD with or without PMS.

DETAILED DESCRIPTION:
Using a non-invasive, pain-free, taste-based approach to assess lidocaine effectiveness, the study will assess the frequency of ineffectiveness in the target population. We will use an identical protocol at two sites: Jacobi hospital and Boston Clinical Trials.

The controlled trial will assess the ability of lidocaine oral gel to block taste (e.g., sweet) in 100 teens and adults, half with a history of ADHD, and for females, we will compare the sub-groups with and without premenstrual syndrome (PMS).

This study will also be compared with a similar assessment among a specialized ADHD population (NCT03563573), that does not respond to existing medication..

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria for both arms:

(1) known adverse reactions to lidocaine; (2) ADHD, ADD, and other inattention disorders; (3) epilepsy, IQ <80, severe head trauma, birth weight <2270 grams, and severe autism; (4) treatment currently with potassium or potassium-elevating drugs such as renin-angiotensin-aldosterone blockers; (5) generalized anxiety disorders (but dental-specific anxiety will not be an exclusion because many of these individuals may be ones with anxiety because of painful dental experiences with lidocaine ineffectiveness); (6) mouth sores; (7) Ehlers Danlos syndrome, (8) red hair, and (9) current pregnancy.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Segal, MD PhD, Principal Investigator — PhenoSolve, LLC
Locations (2):
- United States (2):
  - Boston Clinical Trials, Boston, Massachusetts
  - Jacobi Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
We plan to submit for publication descriptions of what was accomplished, and the evaluations as described in the study, including the incidence of lidocaine ineffectiveness in those with ADHD and in the general population.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 9-12 months
Access Criteria: Researchers
URL: https://phenosolve.com

REFERENCES:
- [Background] Infante MA, Moore EM, Nguyen TT, Fourligas N, Mattson SN, Riley EP. Objective assessment of ADHD core symptoms in children with heavy prenatal alcohol exposure. Physiol Behav. 2015 Sep 1;148:45-50. doi: 10.1016/j.physbeh.2014.10.014. Epub 2014 Oct 23. PMID 25447751
- [Background] Levitt JO. Practical aspects in the management of hypokalemic periodic paralysis. J Transl Med. 2008 Apr 21;6:18. doi: 10.1186/1479-5876-6-18. PMID 18426576
- [Background] Nakai Y, Milgrom P, Mancl L, Coldwell SE, Domoto PK, Ramsay DS. Effectiveness of local anesthesia in pediatric dental practice. J Am Dent Assoc. 2000 Dec;131(12):1699-705. doi: 10.14219/jada.archive.2000.0115. PMID 11143733
- [Background] Segal MM. We cannot say whether attention deficit hyperactivity disorder exists, but we can find its molecular mechanisms. Pediatr Neurol. 2014 Jul;51(1):15-6. doi: 10.1016/j.pediatrneurol.2014.04.014. Epub 2014 Apr 18. No abstract available. PMID 24938135
- [Background] Segal MM, Rogers GF, Needleman HL, Chapman CA. Hypokalemic sensory overstimulation. J Child Neurol. 2007 Dec;22(12):1408-10. doi: 10.1177/0883073807307095. PMID 18174562
- [Background] Segal MM, Douglas AF. Late sodium channel openings underlying epileptiform activity are preferentially diminished by the anticonvulsant phenytoin. J Neurophysiol. 1997 Jun;77(6):3021-34. doi: 10.1152/jn.1997.77.6.3021. PMID 9212254
- [Background] Teicher MH, Polcari A, Fourligas N, Vitaliano G, Navalta CP. Hyperactivity persists in male and female adults with ADHD and remains a highly discriminative feature of the disorder: a case-control study. BMC Psychiatry. 2012 Nov 7;12:190. doi: 10.1186/1471-244X-12-190. PMID 23134619
- See also: Saul R (2014) "ADHD Does Not Exist". HarperCollins — https://www.amazon.com/ADHD-Does-Not-Exist-Hyperactivity/dp/006226673X
- See also: Rozanski RJ, Primosch RE, Courts FJ (1988). Clinical efficacy of 1 and 2% solutions of lidocaine. Pediatr Dent.10:287-90 — https://pdfs.semanticscholar.org/1778/f693dc7dd257ab98a96b5bf03408d9cef3eb.pdf
- See also: Segal MM, Jurkat-Rott K, Levitt J, Lehmann-Horn F (2014) Hypokalemic periodic paralysis - an owner's manual — https://www.uni-ulm.de/fileadmin/website_uni_ulm/med.inst.040/Dokumente/owner.html
- See also: Segal MM (2015) Devices, Kits, and Methods for Determining Sensitivity to Anesthetics. US Patent Filing 62/210,747, Filed 09/14/2015 — https://patents.google.com/patent/WO2017035470A1/en
- See also: Companion study — https://clinicaltrials.gov/ct2/show/NCT03563573

RESULTS

PARTICIPANT FLOW:
Groups:
- Males Without ADHD: Arm 1
  Lidocaine gel: Lidocaine gel 5%
- Males With ADHD: Arm 2
  Lidocaine gel: Lidocaine gel 5%
- Females Without ADHD and Without PMS: Arm 3
  Lidocaine gel: Lidocaine gel 5%
- Females Without ADHD, But With PMS: Arm 4
  Lidocaine gel: Lidocaine gel 5%
- Females With ADHD and Without PMS: Arm 5
  Lidocaine gel: Lidocaine gel 5%
- Females With ADHD and With PMS: Arm 6
  Lidocaine gel: Lidocaine gel 5%
Period: Overall Study
Arm/Group | Males Without ADHD | Males With ADHD | Females Without ADHD and Without PMS | Females Without ADHD, But With PMS | Females With ADHD and Without PMS | Females With ADHD and With PMS
Started | 23 | 14 | 22 | 5 | 15 | 11
Completed | 23 | 14 | 22 | 5 | 15 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Males Without ADHD: ADHD-RS <18
- Males With ADHD: ADHD-RS ≥18
- Females Without ADHD and Without PMS: ADHD-RS <18 and Custom PMS <12
- Females Without ADHD, But With PMS: ADHD-RS <18 and Custom PMS ≥12
- Females With ADHD and Without PMS: ADHD-RS ≥18 and Custom PMS <12
- Females With ADHD and With PMS: ADHD-RS ≥18 and Custom PMS ≥12
- Total: Total of all reporting groups
Arm/Group | Males Without ADHD | Males With ADHD | Females Without ADHD and Without PMS | Females Without ADHD, But With PMS | Females With ADHD and Without PMS | Females With ADHD and With PMS | Total
Number analyzed (Participants) | 23 | 14 | 22 | 5 | 15 | 11 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 14 | 22 | 5 | 15 | 11 | 90
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (7.6) | 27 (7.1) | 33 (6.4) | 33 (10.0) | 27 (6.1) | 30 (8.1) | 30 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 22 | 5 | 15 | 11 | 53
  Male | 23 | 14 | 0 | 0 | 0 | 0 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 6 | 2 | 4 | 4 | 24
  Not Hispanic or Latino | 18 | 11 | 16 | 3 | 11 | 7 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 1 | 1 | 0 | 2 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 2 | 7 | 1 | 2 | 2 | 22
  White | 7 | 8 | 10 | 4 | 9 | 6 | 44
  More than one race | 3 | 1 | 1 | 0 | 2 | 2 | 9
  Unknown or Not Reported | 3 | 2 | 2 | 0 | 0 | 1 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 14 | 22 | 5 | 15 | 11 | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Lidocaine Ineffectiveness
Description: Subjects will be asked to identify each taste and its intensity on a 0 (no taste) to 10 (very intense) scale before and after application of Lidocaine. Lidocaine effectiveness was quantitated as the reduction or elimination of taste by lidocaine compared to taste scores reported before lidocaine. For each of the four before/after pairs, the change in taste intensity was calculated, a weighted average score was computed. Incorrectly identified tastes were excluded. Scores of a reduction in taste ≥50% were considered to be lidocaine effective.
Time Frame: 30 minute visit, added on to a regular clinic visit
Measure: Count of Participants; unit: Participants
Arm/Group | Males Without ADHD | Males With ADHD | Females Without ADHD and Without PMS | Females Without ADHD, But With PMS | Females With ADHD and Without PMS | Females With ADHD and With PMS
Number analyzed (Participants) | 23 | 14 | 22 | 5 | 15 | 11
Participants
  Lidocaine effective (gets numb) | 11 | 9 | 16 | 5 | 15 | 3
  Lidocaine ineffective (does not get numb) | 12 | 5 | 6 | 0 | 0 | 8
Statistical Analysis 1: Comparison: Females Without ADHD and Without PMS vs Females Without ADHD, But With PMS vs Females With ADHD and Without PMS vs Females With ADHD and With PMS; Women with PMS vs. without PMS; Test type: Superiority; p = 0.017, Fisher Exact; Odds Ratio (OR) = 5.17
Statistical Analysis 2: Comparison: Females Without ADHD and Without PMS vs Females Without ADHD, But With PMS vs Females With ADHD and Without PMS vs Females With ADHD and With PMS; Women with PMS and with ADHD vs. other women; Test type: Superiority; p = 0.001, Fisher Exact; Odds Ratio (OR) = 16.0
Statistical Analysis 3: Comparison: Males Without ADHD vs Males With ADHD vs Females Without ADHD and Without PMS vs Females Without ADHD, But With PMS vs Females With ADHD and Without PMS vs Females With ADHD and With PMS; ADHD vs. no ADHD; Test type: Superiority; p = 0.8, Fisher Exact; Odds Ratio (OR) = 0.86

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- All Subjects: All subjects were monitored as a single group for adverse reactions
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT03676725/Prot_SAP_000.pdf